CLINICAL TRIAL: NCT00184717
Title: GHLIQUID-1516: A 104-week, Multi-centre, Randomised, Double-blind, Parallel-group, no Treatment Controlled (Open-label) Trial Investigating the Efficacy and Safety of Two Doses of NN-220 in Subjects With Short Stature Born Small for Gestational Age / GHLIQUID-1517: A Long-term, Multi-centre, Randomised, Controlled, Double-blind, Parallel-group Trial, Investigating the Efficacy and Safety of Two Doses of NN-220 in Subjects With Short Stature Born Small for Gestational Age
Brief Title: Growth Hormone Treatment in Children Born Small for Gestational Age (SGA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GHLIQUID-1517; JapicCTI-050137 (Registry Identifier: JAPIC); JapicCTI-050132 (Registry Identifier: JAPIC); 2017-000914-47 (Registry Identifier: EudraCT); NCT00184704 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Foetal Growth Problem; Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 0.033 mg / NN-220 (Experimental): In the 156-week main period, subjects received 0.033 mg/kg/day somatropin (NN-220) s.c. (under the skin) injected at bedtime followed by a 104-week extension period where subjects received 0.033 mg/kg/day somatropin (NN-220) s.c. (under the skin) injected at bedtime
  Interventions: Drug: somatropin
- 0.067 mg / NN-220 (Experimental): In the 156-week main period, subjects received 0.067 mg/kg/day somatropin (NN-220) s.c. (under the skin) injected at bedtime followed by a 104-week extension period where subjects received 0.067 mg/kg/day somatropin (NN-220) s.c. (under the skin) injected at bedtime
  Interventions: Drug: somatropin
- No treatment (No Intervention): No somatropin (NN-220) treatment was given in the 52-week main period. Subjects was re-randomised to recive two dosing regimens (0.033 mg/kg/day or 0.067 mg/kg/day) in the 208-week extension period
- No treatment --> 0.033 mg (Experimental): In the 208-week extension period, subjects received 0.033 mg/kg/day somatropin (NN-220) s.c. (under the skin) injected at bedtime after having received no somatromin (NN-220) treatment in the 52-week main period
  Interventions: Drug: somatropin
- No treatment --> 0.067 mg (Experimental): In the 208-week extension period, subjects received 0.067 mg/kg/day somatropin (NN-220) s.c. (under the skin) injected at bedtime after having received no somatromin (NN-220) treatment in the 52-week main period
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — 0.033 mg/kg/day of NN-220 for s.c. injection in cartridge
  Arms: 0.033 mg / NN-220; No treatment --> 0.033 mg
Drug: somatropin — 0.067 mg/kg/day of NN-220 for s.c. injection in cartridge
  Arms: 0.067 mg / NN-220; No treatment --> 0.067 mg

SUMMARY:
This study is conducted in Japan. The aim of this trial is to assess the efficacy and safety of somatropin in children born small for gestational age (SGA) in Japan.

In the main period, subjects will receive either active treatment for 104 weeks (two dosing regimens) or no treatment for 52 weeks followed by an extension period where subjects who received active treatment for 104 weeks (two years) will continue with the same treatment for further 156 weeks (three years) while those subjects who received no treatment for 52 weeks (one year) will be randomised to receive two dosing regimens for 208 weeks (four years). In total, subjects participate in trial for 260 weeks (five years).

Main period is registered internally at Novo Nordisk as GHLIQUID-1516 while the extension period is registered as GHLIQUID-1517.

ELIGIBILITY:
Inclusion Criteria:

* For MAIN period (GHLIQUID-1516):
* Born small for gestational age (SGA) with birth weight and birth length below the 10th percentile for gestational age, and additional either birth length below or equal to -2.0 standard deviation score (SDS) or birth weight below or equal to -2.0 SDS for gestational age
* Growth failure with height at -2.0 SDS or below for chronological age (CA)
* Normal growth hormone (GH) production, defined as peak GH level > 10 ng/mL in one GH provocation test
* For EXTENSION period (GHLIQUID-1517):
* Subjects who completed the main period
* Chronological age (CA) for boys at least 4 years, but maximum 11 years
* Chronological age (CA) for girls at least 4 years, but maximum 10 years

Exclusion Criteria:

* Subjects with diabetes mellitus
* Subjects suffering from malignancy
* Several medical conditions

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2004-08-18 (Actual); Primary Completion 2006-03-29 (Actual); Study Completion 2009-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Tanaka T, Yokoya S, Seino Y, Togari H, Mishina J, Kappelgaard AM, Fujieda K. Long-term efficacy and safety of two doses of growth hormone in short Japanese children born small for gestational age. Horm Res Paediatr. 2011;76(6):411-8. doi: 10.1159/000334152. Epub 2011 Nov 29. PMID 22156542
- [Result] Kappelgaard AM, Kiyomi F, Horikawa R, Yokoya S, Tanaka T. The impact of long-term growth hormone treatment on metabolic parameters in Japanese patients with short stature born small for gestational age. Horm Res Paediatr. 2014;81(4):272-9. doi: 10.1159/000358196. Epub 2014 Feb 11. PMID 24526136
- [Derived] Horikawa R, Tanaka T, Nishinaga H, Ogawa Y, Yokoya S. The influence of a long-term growth hormone treatment on lipid and glucose metabolism: a randomized trial in short Japanese children born small for gestational age. Int J Pediatr Endocrinol. 2016;2016:19. doi: 10.1186/s13633-016-0036-4. Epub 2016 Oct 26. PMID 27799945
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 44 sites in Japan
Pre-assignment Details: Subjects completed the main period and were offered to continue in the extension period.
Period: Main Period (GHLIQUID-1516)
Arm/Group | 0.033 mg / NN-220 | 0.067 mg / NN-220 | No Treatment | No Treatment --> 0.033 mg | No Treatment --> 0.067 mg
Started | 39 | 38 | 21 | 0 | 0
Exposed to Trial Drug | 38 | 38 | 21 | 0 | 0
Completed | 36 | 36 | 20 | 0 | 0
Not Completed | 3 | 2 | 1 | 0 | 0
Period: Extension Period (GHLIQUID-1517)
Arm/Group | 0.033 mg / NN-220 | 0.067 mg / NN-220 | No Treatment | No Treatment --> 0.033 mg | No Treatment --> 0.067 mg
Started | 33 (Three subjects did not continue in extension period) | 33 (Three subjects did not continue in extension period) | 0 (Re-randomised to receive 0.033 or 0.067 mg) | 10 (Re-randomised from No treatment group) | 10 (Re-randomised from No treatment group)
Completed | 23 | 27 | 0 | 7 | 5
Not Completed | 10 | 6 | 0 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.033 mg / NN-220 | 0.067 mg / NN-220 | No Treatment | Total
Number analyzed (Participants) | 35 | 34 | 15 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.46 (1.37) | 5.15 (1.2) | 5.09 (1.37) | 5.27 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 8 | 33
  Male | 24 | 20 | 7 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 34 | 15 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 35 | 34 | 15 | 84
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 35 | 34 | 15 | 84
Height [Mean (Standard Deviation); unit: cm] | 96.19 (8.48) | 94.57 (7.28) | 94.42 (8.48) | 95.22 (7.96)
Body weight [Mean (Standard Deviation); unit: kg] | 13.31 (2.55) | 12.62 (1.81) | 12.47 (2.93) | 12.88 (2.36)

OUTCOME MEASURES:

1. Primary Outcome: Change in Height Standard Deviation Score (SDS) for Chronological Age (CA) at Week 260 - Subjects Received NN220 Treatment for 5 Years
Description: Height SDS for chronological age were derived as follow; {Height - mean (age, sex)}/ SD (age, sex), where mean (age, sex) and SD (age, sex) were mean and SD of height for corresponding chronological age and sex (data of those in 2000). Height SDS was calculated using mean of three height observations at corresponding visit
Time Frame: Week 0, week 260
Population: Endpoint Analysis Set (EAS) consisted of subjects who participated in GHLIQUID-1517 in the Full Analysis Set (FAS). FAS consisted of subjects who were randomised in each group and have any available efficacy data after receiving NN-220 in GHLIQUID-1516 or GHLIQUID-1517, except subjects with GCP (Good Clinical Practice) nonconformity
Measure: Least Squares Mean (Standard Error); unit: Standard Deviation Score (SDS)
Arm/Group | 0.033 mg / NN-220 | 0.067 mg / NN-220 | No Treatment --> 0.033 mg | No Treatment --> 0.067 mg
Number analyzed (Participants) | 28 | 29 | 0 | 0
Standard Deviation Score (SDS)
  Week 0 | -2.9488 (0.6368) | -2.9047 (0.6718) |  |
  Week 260 | 1.2066 (0.1102) | 2.0247 (0.1083) |  |

2. Primary Outcome: Change in Height Standard Deviation Score (SDS) for Chronological Age (CA) at Week 208 - Subjects Received NN220 Treatment for 4 Years
Description: as for outcome 1
Time Frame: Week 0, week 208
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Standard Deviation Score (SDS)
Arm/Group | 0.033 mg / NN-220 | 0.067 mg / NN-220 | No Treatment --> 0.033 mg | No Treatment --> 0.067 mg
Number analyzed (Participants) | 0 | 0 | 7 | 8
Standard Deviation Score (SDS)
  Week 0 |  |  | -2.9603 (0.6689) | -2.7481 (0.3524)
  Week 208 |  |  | 1.0997 (0.2453) | 1.9151 (0.2275)

3. Secondary Outcome: Yearly Height Velocity SDS for Chronological Age - Subjects Received NN220 Treatment for 5 Years
Description: Yearly Height velocity SDS for chronological age were summarised and graphically presented
Time Frame: Weeks 0-260
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS)
Arm/Group | 0.033 mg / NN-220 | 0.067 mg / NN-220 | No Treatment --> 0.033 mg | No Treatment --> 0.067 mg
Number analyzed (Participants) | 31 | 34 | 0 | 0
Standard Deviation Score (SDS)
  Baseline, n=31, 34 | -1.6299 (0.9738) | -2.0303 (1.4527) |  |
  Week 52, n=29, 34 | 2.4717 (1.9848) | 4.7875 (1.9365) |  |
  Week 104, n=29, 32 | 1.1344 (1.2782) | 2.8877 (1.1272) |  |
  Week 156, n=25, 29 | 0.8015 (1.0583) | 2.1641 (1.5929) |  |
  Week 208, n=25, 28 | 0.3991 (1.3006) | 1.4724 (1.8696) |  |
  Week 260, n=23, 27 | 0.4612 (2.1558) | 0.7973 (2.1822) |  |

4. Secondary Outcome: Yearly Height Velocity SDS for Chronological Age - Subjects Received NN220 Treatment for 4 Years
Description: Yearly Height velocity SDS for chronological age were summarised and graphically presented
Time Frame: Weeks 0-208
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS)
Arm/Group | 0.033 mg / NN-220 | 0.067 mg / NN-220 | No Treatment --> 0.033 mg | No Treatment --> 0.067 mg
Number analyzed (Participants) | 0 | 0 | 7 | 8
Standard Deviation Score (SDS)
  Baseline, n=7,8 |  |  | 0.073 (1.5681) | -1.356 (0.708)
  Week 52, n=7, 8 |  |  | 2.1677 (0.61) | 5.9303 (1.2096)
  Week 104, n=6, 7 |  |  | 1.5268 (1.1715) | 3.3979 (1.0542)
  Week 156, n=6, 7 |  |  | 1.7617 (2.0956) | 2.3539 (1.3149)
  Week 208, n=6, 6 |  |  | 0.5475 (1.6055) | 2.199 (1.5973)

5. Secondary Outcome: Change in Bone Age (Left Hand X-Ray) at Week 260 - Subjects Received NN220 Treatment for 5 Years
Description: Bone age is measured as years and months (displayed as xx.x years). Change in Bone age = Bone age at 52*i weeks - Bone age at 52*(i-1) weeks, i=1, 2, ….
Time Frame: Week 0, week 260
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: years
Arm/Group | 0.033 mg / NN-220 | 0.067 mg / NN-220 | No Treatment --> 0.033 mg | No Treatment --> 0.067 mg
Number analyzed (Participants) | 21 | 26 | 0 | 0
years | 5.79 (1.05) | 7.15 (1.05) |  |

6. Secondary Outcome: Change in Bone Age (Left Hand X-Ray) at Week 208 - Subjects Received NN220 Treatment for 4 Years
Description: Bone age is measured as years and months (displayed as xx.x years).Change in Bone age = Bone age at 52*i weeks - Bone age at 52*(i-1) weeks, i=1, 2, ….
Time Frame: Week 0, week 208
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: years
Arm/Group | 0.033 mg / NN-220 | 0.067 mg / NN-220 | No Treatment --> 0.033 mg | No Treatment --> 0.067 mg
Number analyzed (Participants) | 0 | 0 | 5 | 6
years |  |  | 6.54 (1.26) | 5.6 (1.68)

7. Secondary Outcome: Adverse Events - Subjects Received NN220 Treatment for 5 Years
Description: Occurrence of Adverse Events (AEs) during treatment period (TEAEs), occurrence of possibly/probably related AEs during the treatment period, and occurrence of Serious Adverse Events (SAEs) during the treatment period. An AE is any undesirable medical event occurring to a subject in a clinical trial, whether or not related to the trial product(s). An SAE is an experience that at any dose is fatal, life-threatening, disabling or which results in the patient being hospitalised or, if already in hospital, that hospitalisation is prolonged, or ocurrence of congenital anomaly
Time Frame: Weeks 0-260
Population: Safety analysis set consisted of all subjects who received at least one dose of NN-220 in GHLIQUID-1516 or GHLIQUID-1517, except subjects with GCP (Good Clinical Practice) nonconformity
Measure: Number; unit: Subjects
Arm/Group | 0.033 mg / NN-220 | 0.067 mg / NN-220 | No Treatment --> 0.033 mg | No Treatment --> 0.067 mg
Number analyzed (Participants) | 31 | 34 | 0 | 0
Subjects
  AEs | 31 | 34 |  |
  AEs possibly/probably related | 9 | 16 |  |
  SAEs | 2 | 4 |  |

8. Secondary Outcome: Adverse Events - Subjects Received NN220 Treatment for 4 Years
Description: as for outcome 7
Time Frame: Weeks 0-208
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | 0.033 mg / NN-220 | 0.067 mg / NN-220 | No Treatment --> 0.033 mg | No Treatment --> 0.067 mg
Number analyzed (Participants) | 0 | 0 | 7 | 8
Subjects
  AEs |  |  | 7 | 8
  AEs possibly/probably relate |  |  | 1 | 3
  SAEs |  |  | 0 | 1

ADVERSE EVENTS:
Time Frame: The adverse events were collected from Aug 2004 to Dec 2009.
Description: The safety analysis set consisted of all subjects who received at least one dose of NN-220 in GHLIQUID-1516 or GHLIQUID-1517, except subjects with GCP nonconformity.
Arm/Group | 0.033 mg / NN-220 | 0.067 mg / NN-220 | 0.033 mg / No Treatment | 0.067 mg / No Treatment
Serious Adverse Events (participants affected / at risk) | 12/31 | 11/34 | 1/7 | 2/8
Other Adverse Events (participants affected / at risk) | 31/31 | 34/34 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.033 mg / NN-220 (N=31) | 0.067 mg / NN-220 (N=34) | 0.033 mg / No Treatment (N=7) | 0.067 mg / No Treatment (N=8)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mumps (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sebaceous naevus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Strabismus (Eye disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular retraction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.033 mg / NN-220 (N=31) | 0.067 mg / NN-220 (N=34) | 0.033 mg / No Treatment (N=7) | 0.067 mg / No Treatment (N=8)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (3) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 2 (8) | 0 (0) | 1 (2)
Acute tonsillitis (Infections and infestations) | 2 (2) | 4 (11) | 0 (0) | 0 (0)
Adenoviral conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Antibody test positive (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 6 (10) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (2) | 2 (2) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 5 (26) | 1 (1) | 2 (2)
Astigmatism (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 4 (5) | 4 (5) | 0 (0) | 1 (2)
Blood urine present (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 14 (66) | 15 (66) | 0 (0) | 6 (19)
Chillblains (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 4 (4) | 7 (13) | 0 (0) | 3 (4)
Conjunctivitis allergic (Eye disorders) | 3 (5) | 5 (7) | 0 (0) | 2 (3)
Constipation (Gastrointestinal disorders) | 6 (8) | 5 (7) | 0 (0) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 6 (7) | 0 (0) | 2 (2)
Convulsion (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (7) | 1 (1) | 1 (1)
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 2 (2) | 6 (7) | 0 (0) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 4 (5) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 9 (14) | 10 (24) | 2 (2) | 2 (2)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Enterobiasis (Infections and infestations) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (8) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis viral (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Enuresis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Febrile convulsion (Nervous system disorders) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Fibromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 10 (18) | 14 (25) | 0 (0) | 1 (2)
Gastroenteritis viral (Infections and infestations) | 11 (20) | 9 (14) | 0 (0) | 4 (8)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 4 (10) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (2) | 2 (2) | 0 (0) | 2 (4)
Herpes simplex (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 6 (9) | 9 (9) | 2 (5) | 1 (2)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 16 (30) | 25 (39) | 6 (7) | 4 (7)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Lymphadenitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (5) | 2 (2) | 0 (0) | 0 (0)
Mumps (Infections and infestations) | 5 (5) | 6 (6) | 1 (1) | 1 (1)
Myopia (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 19 (66) | 27 (212) | 6 (38) | 5 (20)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 7 (11) | 12 (17) | 1 (11) | 3 (12)
Otitis media acute (Infections and infestations) | 4 (13) | 4 (6) | 1 (1) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (7) | 1 (1) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 8 (46) | 14 (74) | 2 (8) | 3 (9)
Pneumonia mycoplasmal (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 10 (17) | 10 (23) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 5 (9) | 6 (9) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 8 (21) | 1 (1) | 5 (6)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (4) | 0 (0) | 1 (4)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 5 (9) | 1 (1) | 1 (9)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (4) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Strabismus (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 7 (19) | 1 (1) | 2 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 22 (147) | 22 (94) | 5 (14) | 6 (32)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 6 (6) | 4 (4) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7) | 4 (6) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk acknowledges the Investigator's right to publish the entire results of the trial. Any such scientific paper, presentation, communication or other information concerning the investigation described in this protocol, must be submitted in writing to Novo Nordisk Trial Manager prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.